CLINICAL TRIAL: NCT00799617
Title: Randomized, Placebo-controlled, Double-blind Study of Seven Coordinated Testosterone Treatment Trials in Older Men
Brief Title: The Testosterone Trials in Older Men
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Aging (NIA) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: U01AG030644 (NIH); R01AG037679 (NIH)
Record Dates: First submitted 2008-11-26; First posted 2008-12-01 (Estimated); Results first posted 2017-08-28 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Andropause
Keywords: Testosterone; Mobility disability; Decreased libido; Age associated memory impairment; Low vitality; Anemia
MeSH Terms: conditions — Anemia | interventions — Testosterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AndroGel® (testosterone gel) (Active Comparator): The initial dose of AndroGel will be 5.0 g (containing 50 mg of testosterone) once a day. Participants will apply AndroGel once daily to the shoulders, abdomen or upper arms. The serum testosterone concentration will be measured monthly for the first three months, then at months 6, 9 and 12. If the testosterone concentration is not between 500 and 800 ng/dL at any time point, the dose will be either increased by increments of 1.25-2.5 g/day, up to a maximum of 15 g/day or decreased by increments of 1.25-3.75 ng/day. Participants will be taught how to apply the gel and they will be provided with written instructions and precautions. This information will be reviewed at each contact and visit.
  Interventions: Drug: AndroGel® (testosterone gel)
- Placebo gel (Placebo Comparator): Placebo gel is identical to the testosterone gel and is supplied in an identical pump bottle container. It is applied to the shoulders, abdomen or upper arms once a day. Participants will be taught how to apply the gel and they will be provided with written instructions and precautions. This information will be reviewed at each contact and visit.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AndroGel® (testosterone gel) — Testosterone levels will be measured at regular intervals in order to achieve a testosterone level in the desired range.
  Other Names: Testosterone gel
  Arms: AndroGel® (testosterone gel)
Drug: Placebo — Testosterone levels will be measured at regular intervals.
  Arms: Placebo gel

SUMMARY:
The Testosterone Trials are a multi-center set of trials involving 12 clinical sites geographically distributed across the United States.

The primary specific aims are to test the hypotheses that testosterone treatment of elderly men whose serum testosterone concentrations are unequivocally low - and who have symptoms and objectively measured abnormalities in at least one of five areas that could be due to low testosterone (physical or sexual function, vitality, cognition, and anemia) - will result in more favorable changes in those abnormalities than placebo treatment.

Two additional trials have been incorporated into the T Trial. Only men enrolled in the T Trial are eligible to participate in these trials.

* The Cardiovascular Trial will examine if testosterone treatment results in more favorable changes in cardiovascular risk factors, compared to placebo.
* The Bone Trial will test the hypothesis that testosterone treatment will increase volumetric trabecular bone mineral density (vBMD) of the lumbar spine as measured by quantitative computed tomography (QCT), compared with placebo treatment.

A Pharmacokinetic (PK) Study is also being conducted within the context of the interventional T Trial. It will examine the variability of the serum testosterone (T) concentration after application of testosterone gel or placebo, four months after the start of treatment.

DETAILED DESCRIPTION:
As men get older, they experience many conditions, often together, that eventually result in the inability to perform many activities of daily living, an increased propensity to fall, and decreased independence. These conditions include mobility disability and low vitality. Elderly men also experience increased anemia, metabolic syndrome, decreased sexual function and memory impairment. These conditions likely have multiple causes, but one cause that could contribute to all of them is a low serum testosterone concentration. When young hypogonadal men are treated with testosterone, they experience improvements in sexual function, muscle mass and strength, bone mineral density, sense of well being, and anemia. However, the benefits of testosterone therapy in older men with age-related decline in testosterone concentration are not known and are the subject of this investigation.

Participants will be treated with testosterone or placebo gel for 1 year. The dose will be adjusted in a blinded fashion to achieve a target T level range. Participants will be followed for one additional year following the treatment phase to assess adverse events.

* Men participating in the Cardiovascular Trial will be assessed for changes in atherosclerotic plaque burden from 0 to 12 months.
* Men participating in the Bone Trial will be assessed by QCT of the spine and hip, DXA of the spine and hip and clinical fractures at 0 and 12 months.
* Men participating in the PK Study will attend 3 additional study visits for blood draws at the time of the 4-month assessment.

ELIGIBILITY:
Inclusion Criteria:

* Men greater than or equal to 65 years old
* Total serum testosterone concentration < 275 and < 300 ng/dL at 7 -10 AM at each of two screening visits

Exclusion Criteria:

* Diagnosed prostate cancer, prostatic intraepithelial neoplasia (PIN), prostate nodule or, by the Prostate Cancer Risk Calculator, a >35% risk of having overall prostate cancer or >7% risk of having high grade prostate cancer
* Severe lower urinary tract symptoms (score of > 19) by the International Prostate Symptom Score questionnaire
* Hemoglobin <10 g/dL or >16.0 g/dL
* Sleep apnea, diagnosed but untreated
* Alcohol or substance abuse within the past year (based on self report)
* Angina not controlled by treatment
* NYHA class III or IV congestive heart failure
* Myocardial infarction within the previous 3 months before entry
* Stroke within the previous 3 months before entry
* Severe pulmonary disease that precludes physical function tests
* Serum creatinine >2.2 mg/dL; ALT 3x upper limit of normal; hemoglobin A1c >8.5%, TSH > 7.5mIU/L
* Diagnosis or treatment for cancer within the past 3 years, with the exception of nonmelanotic skin cancer
* Body mass index (BMI) >37 kg/m2
* Mini Mental State Exam (MMSE) Score <24
* Major psychiatric disorders, including major depression (PHQ-9 score > 14), mania, hypomania, psychosis, schizophrenia or schizoaffective disorders, that are untreated, unstable, have resulted in hospitalization or medication change within the previous three months, or would result in inability to complete the trial efficacy instruments. Subjects whose disorders have been stable while being treated for more than three months are eligible.
* Use of the following medications within the previous three months:

  * drugs that affect serum testosterone concentration
  * rhGH or megestrol acetate
  * introduction of anti-depressant medication
  * daily use of prednisone for more than two weeks
* Opiate use within the past three months
* Skin conditions at the testosterone gel application site, such as ulcer, erosion, lichenification, inflammation, or crust, or generalized skin conditions such as psoriasis or eczema that might affect testosterone absorption or tolerability of the testosterone gel
* Known skin intolerance to alcohol or allergy to any of the ingredients of testosterone gel

Participants in the T Trial may also enroll in the Cardiovascular and Bone Trials if it is determined that they are eligible based on the specific exclusion criteria.

Min Age: 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 790 (Actual)
Dates: Start 2009-11; Primary Completion 2014-07 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Snyder, MD, Principal Investigator — University of Pennsylvania
Locations (12):
- United States (12):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California San Diego, La Jolla, California
  - Center for Men's Health LA BioMed at Harbor-UCLA Medical Center, Torrance, California
  - Yale University, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - Northwestern University, Chicago, Illinois
  - Boston University, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Albert Einstein College of Medicine, The Bronx, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - VA Puget Sound Health Care System, Seattle, Washington

REFERENCES:
- [Derived] Lee H, Hwang EC, Oh CK, Lee S, Yu HS, Lim JS, Kim HW, Walsh T, Kim MH, Jung JH, Dahm P. Testosterone replacement in men with sexual dysfunction. Cochrane Database Syst Rev. 2024 Jan 15;1(1):CD013071. doi: 10.1002/14651858.CD013071.pub2. PMID 38224135
- [Derived] Stephens-Shields AJ, Snyder PJ, Ellenberg SS, Taylor L, Bhasin S. Relation of Testosterone, Dihydrotestosterone, and Estradiol With Changes in Outcomes Measures in the Testosterone Trials. J Clin Endocrinol Metab. 2022 Apr 19;107(5):1257-1269. doi: 10.1210/clinem/dgac028. PMID 35041751
- [Derived] Artz AS, Stephens-Shields AJ, Bhasin S, Ellenberg SS, Cohen HJ, Snyder PJ. Markers of Iron Flux during Testosterone-Mediated Erythropoiesis in Older Men with Unexplained or Iron-Deficiency Anemia. J Clin Endocrinol Metab. 2020 Nov 1;105(11):3396-403. doi: 10.1210/clinem/dgaa521. PMID 32785689
- [Derived] Shaikh K, Ellenberg SS, Nakanishi R, Snyder PJ, Lee J, Wenger NK, Lewis CE, Swerdloff RS, Preston P, Hamal S, Stephens-Sheilds A, Bhasin S, Cherukuri L, Cauley JA, Crandall JP, Cunningham GR, Ensrud KE, Matsumoto AM, Molich ME, Alla VM, Birudaraju D, Nezarat N, Rai K, Almeida S, Roy SK, Sheikh M, Trad G, Budoff MJ. Biomarkers and Noncalcified Coronary Artery Plaque Progression in Older Men Treated With Testosterone. J Clin Endocrinol Metab. 2020 Jul 1;105(7):2142-9. doi: 10.1210/clinem/dgz242. PMID 31784747
- [Derived] Bhasin S, Ellenberg SS, Storer TW, Basaria S, Pahor M, Stephens-Shields AJ, Cauley JA, Ensrud KE, Farrar JT, Cella D, Matsumoto AM, Cunningham GR, Swerdloff RS, Wang C, Lewis CE, Molitch ME, Barrett-Connor E, Crandall JP, Hou X, Preston P, Cifelli D, Snyder PJ, Gill TM. Effect of testosterone replacement on measures of mobility in older men with mobility limitation and low testosterone concentrations: secondary analyses of the Testosterone Trials. Lancet Diabetes Endocrinol. 2018 Nov;6(11):879-890. doi: 10.1016/S2213-8587(18)30171-2. PMID 30366567
- [Derived] Mohler ER 3rd, Ellenberg SS, Lewis CE, Wenger NK, Budoff MJ, Lewis MR, Barrett-Connor E, Swerdloff RS, Stephens-Shields A, Bhasin S, Cauley JA, Crandall JP, Cunningham GR, Ensrud KE, Gill TM, Matsumoto AM, Molitch ME, Pahor M, Preston PE, Hou X, Cifelli D, Snyder PJ. The Effect of Testosterone on Cardiovascular Biomarkers in the Testosterone Trials. J Clin Endocrinol Metab. 2018 Feb 1;103(2):681-688. doi: 10.1210/jc.2017-02243. PMID 29253154
- [Derived] Resnick SM, Matsumoto AM, Stephens-Shields AJ, Ellenberg SS, Gill TM, Shumaker SA, Pleasants DD, Barrett-Connor E, Bhasin S, Cauley JA, Cella D, Crandall JP, Cunningham GR, Ensrud KE, Farrar JT, Lewis CE, Molitch ME, Pahor M, Swerdloff RS, Cifelli D, Anton S, Basaria S, Diem SJ, Wang C, Hou X, Snyder PJ. Testosterone Treatment and Cognitive Function in Older Men With Low Testosterone and Age-Associated Memory Impairment. JAMA. 2017 Feb 21;317(7):717-727. doi: 10.1001/jama.2016.21044. PMID 28241356
- [Derived] Budoff MJ, Ellenberg SS, Lewis CE, Mohler ER 3rd, Wenger NK, Bhasin S, Barrett-Connor E, Swerdloff RS, Stephens-Shields A, Cauley JA, Crandall JP, Cunningham GR, Ensrud KE, Gill TM, Matsumoto AM, Molitch ME, Nakanishi R, Nezarat N, Matsumoto S, Hou X, Basaria S, Diem SJ, Wang C, Cifelli D, Snyder PJ. Testosterone Treatment and Coronary Artery Plaque Volume in Older Men With Low Testosterone. JAMA. 2017 Feb 21;317(7):708-716. doi: 10.1001/jama.2016.21043. PMID 28241355
- [Derived] Roy CN, Snyder PJ, Stephens-Shields AJ, Artz AS, Bhasin S, Cohen HJ, Farrar JT, Gill TM, Zeldow B, Cella D, Barrett-Connor E, Cauley JA, Crandall JP, Cunningham GR, Ensrud KE, Lewis CE, Matsumoto AM, Molitch ME, Pahor M, Swerdloff RS, Cifelli D, Hou X, Resnick SM, Walston JD, Anton S, Basaria S, Diem SJ, Wang C, Schrier SL, Ellenberg SS. Association of Testosterone Levels With Anemia in Older Men: A Controlled Clinical Trial. JAMA Intern Med. 2017 Apr 1;177(4):480-490. doi: 10.1001/jamainternmed.2016.9540. PMID 28241237
- [Derived] Snyder PJ, Kopperdahl DL, Stephens-Shields AJ, Ellenberg SS, Cauley JA, Ensrud KE, Lewis CE, Barrett-Connor E, Schwartz AV, Lee DC, Bhasin S, Cunningham GR, Gill TM, Matsumoto AM, Swerdloff RS, Basaria S, Diem SJ, Wang C, Hou X, Cifelli D, Dougar D, Zeldow B, Bauer DC, Keaveny TM. Effect of Testosterone Treatment on Volumetric Bone Density and Strength in Older Men With Low Testosterone: A Controlled Clinical Trial. JAMA Intern Med. 2017 Apr 1;177(4):471-479. doi: 10.1001/jamainternmed.2016.9539. PMID 28241231
- [Derived] Cunningham GR, Stephens-Shields AJ, Rosen RC, Wang C, Bhasin S, Matsumoto AM, Parsons JK, Gill TM, Molitch ME, Farrar JT, Cella D, Barrett-Connor E, Cauley JA, Cifelli D, Crandall JP, Ensrud KE, Gallagher L, Zeldow B, Lewis CE, Pahor M, Swerdloff RS, Hou X, Anton S, Basaria S, Diem SJ, Tabatabaie V, Ellenberg SS, Snyder PJ. Testosterone Treatment and Sexual Function in Older Men With Low Testosterone Levels. J Clin Endocrinol Metab. 2016 Aug;101(8):3096-104. doi: 10.1210/jc.2016-1645. Epub 2016 Jun 29. PMID 27355400
- [Derived] Snyder PJ, Bhasin S, Cunningham GR, Matsumoto AM, Stephens-Shields AJ, Cauley JA, Gill TM, Barrett-Connor E, Swerdloff RS, Wang C, Ensrud KE, Lewis CE, Farrar JT, Cella D, Rosen RC, Pahor M, Crandall JP, Molitch ME, Cifelli D, Dougar D, Fluharty L, Resnick SM, Storer TW, Anton S, Basaria S, Diem SJ, Hou X, Mohler ER 3rd, Parsons JK, Wenger NK, Zeldow B, Landis JR, Ellenberg SS; Testosterone Trials Investigators. Effects of Testosterone Treatment in Older Men. N Engl J Med. 2016 Feb 18;374(7):611-24. doi: 10.1056/NEJMoa1506119. PMID 26886521
- [Derived] Abd Alamir M, Ellenberg SS, Swerdloff RS, Wenger NK, Mohler ER 3rd, Lewis CE, Barrett-Conner E, Nakanishi R, Darabian S, Alani A, Matsumoto S, Nezarat N, Snyder PJ, Budoff MJ. The Cardiovascular Trial of the Testosterone Trials: rationale, design, and baseline data of a clinical trial using computed tomographic imaging to assess the progression of coronary atherosclerosis. Coron Artery Dis. 2016 Mar;27(2):95-103. doi: 10.1097/MCA.0000000000000321. PMID 26554661
- [Derived] Cunningham GR, Stephens-Shields AJ, Rosen RC, Wang C, Ellenberg SS, Matsumoto AM, Bhasin S, Molitch ME, Farrar JT, Cella D, Barrett-Connor E, Cauley JA, Cifelli D, Crandall JP, Ensrud KE, Fluharty L, Gill TM, Lewis CE, Pahor M, Resnick SM, Storer TW, Swerdloff RS, Anton S, Basaria S, Diem S, Tabatabaie V, Hou X, Snyder PJ. Association of sex hormones with sexual function, vitality, and physical function of symptomatic older men with low testosterone levels at baseline in the testosterone trials. J Clin Endocrinol Metab. 2015 Mar;100(3):1146-55. doi: 10.1210/jc.2014-3818. Epub 2014 Dec 30. PMID 25548978
- [Derived] Meng J, Mostaghel EA, Vakar-Lopez F, Montgomery B, True L, Nelson PS. Testosterone regulates tight junction proteins and influences prostatic autoimmune responses. Horm Cancer. 2011 Jun;2(3):145-56. doi: 10.1007/s12672-010-0063-1. PMID 21761342
- See also: Find out more information about The Testosterone Trial and the list of participating clinical sites. — http://www.trial.org

RESULTS

PARTICIPANT FLOW:
Groups:
- AndroGel® (Testosterone Gel): AndroGel is applied to the shoulders, abdomen or upper arms once a day. Subjects will be instructed to wash their hands after application and not to have contact with women or children while the gel is wet. They will also be asked not to bathe or get this area wet for five hours after application. The initial dose of AndroGel will be 5.0 g (containing 50 mg of testosterone) once a day.
  AndroGel® (testosterone gel): Testosterone levels will be measured at regular intervals in order to achieve a testosterone level in the desired range.
- Placebo Gel: Placebo gel is identical to the testosterone gel and is supplied in an identical pump bottle container. It is applied to the shoulders, abdomen or upper arms once a day. Subjects will be instructed to follow the same precautions to avoid contact with others.
  Placebo: Testosterone levels will be measured at regular intervals.
Period: Main Testosterone Trial
Arm/Group | AndroGel® (Testosterone Gel) | Placebo Gel
Started | 395 | 395
Completed (The Testosterone Trials are a coordinated set of 7 trials.) | 376 (Participants qualified for 1 of the 3 main trials (sexual function, physical function, vitality).) | 374
Not Completed | 19 | 21
Not completed — Randomized in error | 1 | 1
Not completed — Lost to Follow-up | 18 | 20
Period: Sexual Funtion Trial
Arm/Group | AndroGel® (Testosterone Gel) | Placebo Gel
Started | 234 | 236
Completed | 218 | 215
Not Completed | 16 | 21
Not completed — Lost to Follow-up | 12 | 14
Not completed — No Baseline Data | 4 | 7
Period: Physical Function Trial
Arm/Group | AndroGel® (Testosterone Gel) | Placebo Gel
Started | 191 | 196
Completed | 185 | 185
Not Completed | 6 | 11
Not completed — Lost to Follow-up | 6 | 11
Period: Vitality Trial
Arm/Group | AndroGel® (Testosterone Gel) | Placebo Gel
Started | 236 | 238
Completed | 229 | 216
Not Completed | 7 | 22
Not completed — Lost to Follow-up | 7 | 22
Period: Cardiovascular Trial
Arm/Group | AndroGel® (Testosterone Gel) | Placebo Gel
Started | 88 | 82
Completed | 73 | 65
Not Completed | 15 | 17
Not completed — Month 12 scan not available | 15 | 15
Not completed — Baseline scan not analyzable | 0 | 2
Period: Bone Trial
Arm/Group | AndroGel® (Testosterone Gel) | Placebo Gel
Started | 110 | 101
Completed | 104 | 85
Not Completed | 6 | 16
Not completed — Month 12 scan not available | 6 | 16
Period: Cognitive Function Trial
Arm/Group | AndroGel® (Testosterone Gel) | Placebo Gel
Started | 247 | 246
Completed | 247 | 245
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Period: Anemia Trial
Arm/Group | AndroGel® (Testosterone Gel) | Placebo Gel
Started | 27 | 35
Completed | 24 | 32
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 3 | 3

BASELINE CHARACTERISTICS:
Population: Two participants were randomized in error, one in each arm of the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | AndroGel® (Testosterone Gel) | Placebo Gel | Total
Number analyzed (Participants) | 394 | 394 | 788
Age, Continuous [Mean (Standard Deviation); unit: years] — Men in the trial were 65 years of age or older. Population: The number analyzed differs from the number randomized because 2 participants were randomized in error. Participants in the Sexual Function, Physical Function and Vitality trials are enrolled in the overall Main Testosterone Trial.
  years
    Main Testosterone Trial | 72.3 (5.8) | 72.1 (5.7) | 72.2 (5.8)
    Cardiovascular Trial: number analyzed (Participants) | 73 | 65 | 138
    Cardiovascular Trial | 70.5 (5.7) | 72.0 (5.7) | 71.2 (5.7)
    Bone Trial: number analyzed (Participants) | 110 | 101 | 211
    Bone Trial | 72.3 (6.3) | 72.4 (5.5) | 72.4 (5.9)
    Cognitive Function Trial: number analyzed (Participants) | 247 | 246 | 493
    Cognitive Function Trial | 72.3 (5.8) | 72.8 (6.1) | 72.6 (5.9)
    Anemia Trial: number analyzed (Participants) | 27 | 35 | 62
    Anemia Trial | 74.8 (6.0) | 75.6 (7.5) | 75.2 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants] — All of the participants in this trial of testosterone gel use are men. Population: The number of participants analyzed differs from the number randomized because some participants withdrew from the trial before month 12 or did not provide complete follow-up data.
  Participants
    Female | 0 | 0 | 0
    Male | 394 | 394 | 788
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 10 | 28
  Not Hispanic or Latino | 375 | 384 | 759
  Unknown or Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian | 348 | 350 | 698
  Race: African-American | 21 | 20 | 41
  Race: Other | 25 | 24 | 49

OUTCOME MEASURES:

1. Primary Outcome: Sexual Function Trial - Change in Psychosexual Daily Questionnaire Question 4 (PDQ-Q4) From Baseline to Month 12
Description: Baseline score and change in responses to Question 4 of the Psychosexual Daily Questionnaire (PDQ-Q4) from baseline to Month 12.
  Question 4 asks 12 questions about sexual activity. Scores on the PDQ-Q4 range from 0 to 12, with higher scores indicating more activity.
  The change is measured form the baseline value to Month 12.
Time Frame: 1 year (change from baseline to month 3, 6, 9 and 12)
Measure: Mean (Standard Deviation); unit: units on the PDQ-Q4 scale
Arm/Group | AndroGel® (Testosterone Gel) | Placebo Gel
Number analyzed (Participants) | 230 | 229
units on the PDQ-Q4 scale
  Baseline Score | 1.4 (1.3) | 1.4 (1.3)
  Change at Month 3 | 0.6 (1.3) | 0.1 (1.1)
  Change at Month 6 | 0.6 (1.5) | -0.1 (1.2)
  Change at Month 9 | 0.5 (1.5) | -0.1 (1.2)
  Change at Month 12 | 0.2 (1.6) | -0.1 (1.4)
Statistical Analysis 1: Comparison: AndroGel® (Testosterone Gel) vs Placebo Gel; Test type: Superiority; p < 0.001, Mixed Models Analysis — The p value for the treatment effect was determined with the use of a linear mixed model with a random effect for participant; Adjustment for balancing factors: baseline testosterone, age, site, trial participation, use of antidepressants, use of PDE5 inhibitors; Mean Difference (Net) = 0.58, 95% CI 2-sided [0.38 to 0.78]

2. Primary Outcome: Physical Function Trial - The 6-Minute Walk Test - no./Total no. (%)
Description: The number and percentage of men who increased the distance walked in the 6-Minute Walk Test by at least 50 meters.
Time Frame: 1 year (Number of participants who increased walk distance > or = 50 meters, change from baseline to month 3, 6, 9 and 12)
Population: The number analyzed differs from the overall number due to participant withdrawal or test results that were incomplete.
Measure: Count of Participants; unit: Participants
Arm/Group | AndroGel® (Testosterone Gel) | Placebo Gel
Number analyzed (Participants) | 191 | 196
Participants
  Month 3: number analyzed (Participants) | 179 | 179
  Month 3 | 20 | 14
  Month 6: number analyzed (Participants) | 174 | 171
  Month 6 | 24 | 23
  Month 9: number analyzed (Participants) | 191 | 159
  Month 9 | 28 | 22
  Month 12 | 35 | 20
Statistical Analysis 1: Comparison: AndroGel® (Testosterone Gel) vs Placebo Gel; The treatment effect for dichotomous outcomes is the odds ratio for achieving the outcome versus not achieving the outcome among men assigned to testosterone versus those assigned to placebo; Test type: Superiority; p = 0.20, Mixed Models Analysis — The P value for the treatment effect was determined with the use of a logistic mixed model with a random effect for participant for dichotomous outcomes and a linear mixed model with a random effect for participant for continuous outcomes; Odds Ratio (OR) = 1.42, 95% CI 2-sided [0.83 to 2.45]

3. Primary Outcome: Vitality Trial - Increase in Functional Assessment of Chronic Illness Therapy (FACIT) - Fatigue Score Greater Than or Equal to 4 - no./Total no. (%)
Description: The number of participants whose score on the FACIT-Fatigue scale increased by at least 4 points.
  Scores on the FACIT- Fatigue scale range from 0 to 52, with higher scores indicating less fatigue.
Time Frame: 1 year (Number of participants who increased FACIT-Fatigue score > or = to 4, change from baseline to month 3, 6, 9 and 12)
Population: The number analyzed differs from the overall number due to participant withdrawal or test results that were incomplete.
Measure: Count of Participants; unit: Participants
Arm/Group | AndroGel® (Testosterone Gel) | Placebo Gel
Number analyzed (Participants) | 236 | 238
Participants
  Month 3: number analyzed (Participants) | 219 | 207
  Month 3 | 148 | 138
  Month 6: number analyzed (Participants) | 217 | 196
  Month 6 | 144 | 126
  Month 9: number analyzed (Participants) | 206 | 188
  Month 9 | 148 | 127
  Month 12 | 147 | 120
Statistical Analysis 1: Comparison: AndroGel® (Testosterone Gel) vs Placebo Gel; Test type: Superiority; p = 0.30, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.83 to 1.84]

4. Primary Outcome: Cardiovascular Trial - Assess Impact of Testosterone Treatment in Older Men on Noncalcified Plaque Volume
Description: Non-calcified coronary artery plaque volume, mm3, as determined by coronary computed tomographic angiography (CTA), mean difference in change from baseline to month 12
Time Frame: 1 year (change in plaque volume measurement from baseline to month 12)
Population: Men aged 65 years or > with an average of 2 serum testosterone levels lower than 275 ng/L and enrolled in the CV Trial of the Testosterone Trials between June 2010 and June 2014.
Measure: Mean (95% Confidence Interval); unit: mm^3
Arm/Group | AndroGel® (Testosterone Gel) | Placebo Gel
Number analyzed (Participants) | 73 | 65
mm^3 | 54 [12 to 97] | 14 [-29 to 56]
Statistical Analysis 1: Comparison: AndroGel® (Testosterone Gel) vs Placebo Gel; Test type: Superiority; p = .003, Regression, Linear — Determined by a linear mixed model with all balancing factors and baseline outcome value as covariates and a random effect for participant; Mean Difference (Final Values) = 41, 95% CI 2-sided [14 to 67] — Mean difference in change from baseline for participants assigned to testosterone v. placebo, with adjustment for balancing factors: baseline testosterone, age, site, trial participation, use of antidepressants, PDE5 inhibitors, baseline outcome

5. Primary Outcome: Bone Trial - Volumetric Bone Mineral Density (BMD) of Spine Trabecular Bone by Quantitative Computed Tomography (QCT) in Older Men With Low Testosterone
Description: Volumetric Bone Mineral Density (BMD) of spine trabecular bone as measured by QCT, mg/cm3, the calculated change in measurement from baseline to Month 12
Time Frame: 1 year (QCT measurement of BMD change between baseline and month 12)
Measure: Mean (95% Confidence Interval); unit: mg/cm^3
Arm/Group | AndroGel® (Testosterone Gel) | Placebo Gel
Number analyzed (Participants) | 110 | 97
mg/cm^3 | 7.5 [4.8 to 10.3] | 0.8 [-1.9 to 3.4]
Statistical Analysis 1: Comparison: AndroGel® (Testosterone Gel) vs Placebo Gel; Test type: Superiority; p < .001, Regression, Linear — Treatment effect is the mean difference in the change from baseline between testosterone and placebo arms.The P-Value for the significance of the treatment effect was determined by multivariable linear regression adjusted for balancing factors; Mean Difference (Final Values) = 6.8, 95% CI 2-sided [4.8 to 8.7]

6. Primary Outcome: Cognitive Function Trial - Delayed Paragraph Recall Wechsler Memory Scale Revised Logical Memory II (WMS-R LMII)
Description: Baseline score and change in score of the Wechsler Memory Scale Revised Logical Memory II (WMS-R LMII) test of Delayed Paragraph Recall, at baseline, Month 6 and Month 12.
  The WMS-R LM II involves a delayed paragraph recall activity scored in two components, each ranging from 0-25. The final score is the sum of each component, therefore falling in the range 0-50. WMS-R LM II scores were treated as continuous with change compared between treatment arms using linear random effects models adjusting for several factors: site, indicator variables of participation in each primary efficacy trial, baseline testosterone concentration (<200), age (≤ 75), use of anti-depressants, use of PDE-inhibitors, baseline WMSR, categorical education, and version of the WMSR.
Time Frame: 1 year (change from baseline to month 6 and month 12)
Population: Men, age 65 years or older with low testosterone and Age-Associated Memory Impairment (AAMI)
Measure: Mean (95% Confidence Interval); unit: percentage of change in test score
Arm/Group | AndroGel® (Testosterone Gel) | Placebo Gel
Number analyzed (Participants) | 247 | 246
percentage of change in test score
  Baseline Score | 14.0 [13.2 to 14.8] | 14.4 [13.6 to 15.2]
  Change at Month 6 | 1.1 [-0.1 to 2.3] | 1.1 [-0.1 to 2.3]
  Change at Month 12 | 1.3 [0.1 to 2.5] | 1.4 [0.3 to 2.6]
Statistical Analysis 1: Comparison: AndroGel® (Testosterone Gel) vs Placebo Gel; A positive estimated difference indicates greater increases, smaller decreases, or both for the testosterone group compared with the placebo group. The difference is the mean difference in the change from baseline to 6 months to 12 months in participants allocated to testosterone vs placebo adjusted for balancing factors; Test type: Superiority; p = .88, Mixed Models Analysis — The estimated difference and P-value were determined by a linear mixed-model with a random effect for participants using outcomes at month 6 and month 12; Mean Difference (Net) = -0.07, 95% CI 2-sided [-0.92 to 0.79]

7. Primary Outcome: Anemia Trial - Effect of Testosterone on Hemoglobin Levels - Unexplained Anemia
Description: Proportion of men age 65 years or older with unexplained anemia who increased their hemoglobin level by 1.0 g/dL from baseline.
  Values are No. (%) for dichotomous outcomes. Dichotomous hemoglobin response is an increase of 1 g/dL or more from baseline.
Time Frame: 1 year (change in hemoglobin g/dL from baseline to month 3, 6, 9 and 12)
Population: Unexplained anemia is anemia that is not due to the following causes: iron and vitamin B12 deficiency, chronic inflammation and disease, chronic renal insufficiency, myelodysplastic syndromes.
Measure: Count of Participants; unit: Participants
Arm/Group | AndroGel® (Testosterone Gel) | Placebo Gel
Number analyzed (Participants) | 27 | 35
Participants
  Month 3: number analyzed (Participants) | 24 | 32
  Month 3 | 6 | 4
  Month 6: number analyzed (Participants) | 22 | 27
  Month 6 | 8 | 3
  Month 9: number analyzed (Participants) | 24 | 28
  Month 9 | 15 | 2
  Month 12: number analyzed (Participants) | 24 | 27
  Month 12 | 13 | 4
Statistical Analysis 1: Comparison: AndroGel® (Testosterone Gel) vs Placebo Gel; Test type: Superiority — Dichotomous hemoglobin response is an increase of 1g/dL or more from baseline; p = .002, Mixed Models Analysis — The P-value for the significance of the treatment effect was determined by a logistic mixed model with a random intercept for participant; The statistical analysis was intent-to-treat by a logistic mixed effects model adjusted for balancing factors; Odds Ratio (OR) = 31.5, 95% CI 2-sided [3.7 to 277.8]

8. Secondary Outcome: Sexual Function Trial - Sexual Desire Domain
Description: Baseline score and the changes in the score of the sexual-desire domain of the Derogatis Interview for Sexual Functioning in Men-II (DISF-M-II), from baseline to Month 12.
  Scores on the (DISF-M-II) range from 0 to 33, with higher scores indicating greater sexual desire.
Time Frame: 1 year (change from baseline to month 3, 6, 9 and 12)
Measure: Mean (Standard Deviation); unit: Score on the DISF-M-II scale
Arm/Group | AndroGel® (Testosterone Gel) | Placebo Gel
Number analyzed (Participants) | 234 | 236
Score on the DISF-M-II scale
  Baseline Score | 11.9 (6.7) | 11.6 (6.6)
  Change at Month 3 | 3.5 (6.3) | 0.7 (5.8)
  Change at Month 6 | 3.5 (6.0) | 0.8 (5.6)
  Change at Month 9 | 4.0 (7.4) | 0.9 (5.5)
  Change at Month 12 | 2.6 (6.5) | 0.0 (5.0)
Statistical Analysis 1: Comparison: AndroGel® (Testosterone Gel) vs Placebo Gel; Test type: Superiority; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 2.93, 95% CI 2-sided [2.13 to 3.74]

9. Secondary Outcome: Sexual Function Trial - Erectile Function
Description: Baseline score and the change in score on the International Index of Erectile Function (IIEF) from baseline to Month 12.
  Scores on the IIEF range from 0-30, with higher scores indicating better function.
Time Frame: 1 year (change from baseline to month 3, 6, 9 and 12)
Measure: Mean (Standard Deviation); unit: Score on the IIEF test scale
Arm/Group | AndroGel® (Testosterone Gel) | Placebo Gel
Number analyzed (Participants) | 234 | 236
Score on the IIEF test scale
  Baseline Score | 8.0 (8.2) | 7.7 (8.2)
  Change at Month 3 | 3.4 (6.1) | 1.0 (5.3)
  Change at Month 6 | 3.3 (6.5) | 0.5 (6.1)
  Change at Month 9 | 3.4 (6.9) | 0.5 (7.1)
  Change at Month 12 | 3.1 (6.9) | 1.0 (6.0)
Statistical Analysis 1: Comparison: AndroGel® (Testosterone Gel) vs Placebo Gel; Test type: Superiority; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Median Difference (Net) = 2.64, 95% CI 2-sided [1.68 to 3.61]

10. Secondary Outcome: Physical Function Trial - 6 Minute Walk Test - Total Walking Distance in Meters
Description: Baseline score and the change in distance walked in the 6-Minute Walking Test in meters from baseline to Month 12
Time Frame: 1 year (change from baseline to month 3, 6, 9 and 12)
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | AndroGel® (Testosterone Gel) | Placebo Gel
Number analyzed (Participants) | 191 | 196
meters
  Baseline Score | 347.7 (69.1) | 344.9 (68.5)
  Change at Month 3 | 10.2 (35.8) | 4.6 (35.2)
  Change at Month 6 | 8.2 (41.5) | 7.8 (41.4)
  Change at Month 9 | 5.3 (50.3) | 3.2 (52.4)
  Change at Month 12 | 14.3 (45.9) | 5.5 (46.4)
Statistical Analysis 1: Comparison: AndroGel® (Testosterone Gel) vs Placebo Gel; Test type: Superiority; p = 0.28, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 4.09, 95% CI 2-sided [-3.00 to 11.18]

11. Secondary Outcome: Physical Function Trial - The Physical Function Domain (PF-10) of the SF-36 - no./Total no. (%)
Description: The number of participants whose score on the physical-function domain (PF-10; range, 0 to 100, with higher scores indicating better function) of the Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36) increased by at least 8 points from baseline to Month 12.
Time Frame: 1 year (change from baseline to month 3, 6, 9 and 12)
Population: The number analyzed differs from the overall number due to participant withdrawal or test results that were incomplete.
Measure: Count of Participants; unit: Participants
Arm/Group | AndroGel® (Testosterone Gel) | Placebo Gel
Number analyzed (Participants) | 184 | 181
Participants
  Month 3: number analyzed (Participants) | 176 | 171
  Month 3 | 77 | 59
  Month 6: number analyzed (Participants) | 171 | 159
  Month 6 | 72 | 73
  Month 9: number analyzed (Participants) | 172 | 159
  Month 9 | 77 | 60
  Month 12 | 66 | 58
Statistical Analysis 1: Comparison: AndroGel® (Testosterone Gel) vs Placebo Gel; Test type: Superiority; p = 0.15, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.34, 95% CI 2-sided [0.90 to 2.00]

12. Secondary Outcome: Physical Function Trial - PF 10 Overall Score
Description: Baseline score and the change in score on the physical-function scale (PF-10) of the Medical Outcomes Study 36-Item Short Form Health Survey range from 0 to 100, with higher scores indicating better function.
  Scores were measured as the change from baseline to Month 12.
Time Frame: 1 year (change from baseline to month 3, 6, 9 and 12)
Measure: Mean (Standard Deviation); unit: Score on the PF-10 test scale
Arm/Group | AndroGel® (Testosterone Gel) | Placebo Gel
Number analyzed (Participants) | 184 | 181
Score on the PF-10 test scale
  Baseline Score | 65.4 (20.0) | 64.8 (21.3)
  Change at Month 3 | 5.6 (15.2) | 4.2 (13.7)
  Change at Month 6 | 6.5 (16.7) | 4.8 (17.0)
  Change at Month 9 | 5.9 (19.4) | 3.3 (18.9)
  Change at Month 12 | 5.8 (17.5) | 2.4 (17.3)
Statistical Analysis 1: Comparison: AndroGel® (Testosterone Gel) vs Placebo Gel; Test type: Superiority; p = 0.03, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 2.75, 95% CI 2-sided [0.20 to 5.29]

13. Secondary Outcome: Vitality Trial - FACIT Fatigue Overall Score
Description: Baseline score and change in the FACIT- Fatigue score from baseline to Month 12. Scores on the Functional Assessment of Chronic Illness Therapy (FACIT) - Fatigue scale range from 0 to 52, with higher scores indicating less fatigue.
Time Frame: 1 year (change from baseline to month 3, 6, 9 and 12)
Measure: Mean (Standard Deviation); unit: Score on the FACIT- Fatigue test scale
Arm/Group | AndroGel® (Testosterone Gel) | Placebo Gel
Number analyzed (Participants) | 236 | 238
Score on the FACIT- Fatigue test scale
  Baseline Score | 31.6 (6.4) | 31.3 (6.4)
  Change at Month 3 | 7.8 (8.4) | 7.2 (8.8)
  Change at Month 6 | 7.4 (9.1) | 5.9 (9.2)
  Change at Month 9 | 8.6 (9.1) | 7.2 (9.2)
  Change at Month 12 | 8.0 (8.4) | 6.7 (9.4)
Statistical Analysis 1: Comparison: AndroGel® (Testosterone Gel) vs Placebo Gel; Test type: Superiority; p = 0.06, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 1.21, 95% CI 2-sided [-0.04 to 2.46]

14. Secondary Outcome: Vitality Trial - SF-36 Score
Description: Baseline score and change in the SF-36 Vitality Score from baseline to Month 12 Scores on the vitality scale of the Medical Outcomes Study 36-Item Short Form Health Survey (SF-36) range from 0 to 100, with higher scores indicating less fatigue.
Time Frame: 1 year (change from baseline to month 3, 6, 9 and 12)
Measure: Mean (Standard Deviation); unit: Score on the SF-36 vitality scale
Arm/Group | AndroGel® (Testosterone Gel) | Placebo Gel
Number analyzed (Participants) | 208 | 196
Score on the SF-36 vitality scale
  Baseline Score | 50.6 (13.8) | 49.4 (12.6)
  Change at Month 3 | 7.4 (13.6) | 5.9 (11.1)
  Change at Month 6 | 7.2 (14.6) | 4.5 (11.2)
  Change at Month 9 | 8.4 (14.4) | 5.7 (12.3)
  Change at Month 12 | 8.2 (15.3) | 6.1 (13.8)
Statistical Analysis 1: Comparison: AndroGel® (Testosterone Gel) vs Placebo Gel; Test type: Superiority or Other; p = 0.03, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 2.41, 95% CI 2-sided [0.31 to 4.50]

15. Secondary Outcome: Vitality Trial - Change in the Positive Affect Score of the Positive and Negative Affect Scales (PANAS) From Baseline to Month 12.
Description: Baseline score and change in the total positive affect score of the Positive and Negative Affect Scales (PANAS) from baseline to Month 12.
  Scores for positive affect and for negative affect on the Positive and Negative Affect Schedule (PANAS) scales range from 5 to 50, with higher scores indicating a greater intensity of the affect.
Time Frame: 1 year (change from baseline to month 3, 6, 9 and 12)
Measure: Mean (Standard Deviation); unit: Score on the PANAS test scale
Arm/Group | AndroGel® (Testosterone Gel) | Placebo Gel
Number analyzed (Participants) | 229 | 234
Score on the PANAS test scale
  Baseline Score | 15.3 (3.2) | 15.4 (3.5)
  Change at Month 3 | 0.7 (3.2) | 0.3 (3.3)
  Change at Month 6 | 0.9 (3.8) | 0.0 (3.3)
  Change at Month 9 | 0.9 (3.4) | 0.4 (3.4)
  Change at Month 12 | 0.7 (3.9) | 0.2 (3.2)
Statistical Analysis 1: Comparison: AndroGel® (Testosterone Gel) vs Placebo Gel; Test type: Superiority or Other; p = 0.04, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 0.47, 95% CI 2-sided [0.02 to 0.92]

16. Secondary Outcome: Vitality Trial - Change in the Total Negative Affect Score of the Positive and Negative Affect Scales (PANAS) From Baseline to Month 12
Description: Baseline score and change in the total negative affect score of the Positive and Negative Affect Scales (PANAS) from baseline to Month 12.
  Scores for positive affect and for negative affect on the Positive and Negative Affect Schedule (PANAS) scales range from 5 to 50, with higher scores indicating a greater intensity of the affect.
Time Frame: 1 year (change from baseline to month 3, 6, 9 and 12)
Measure: Mean (Standard Deviation); unit: Score on the PANAS test scale
Arm/Group | AndroGel® (Testosterone Gel) | Placebo Gel
Number analyzed (Participants) | 229 | 234
Score on the PANAS test scale
  Baseline Score | 7.5 (2.7) | 7.4 (2.8)
  Change at Month 3 | -0.2 (2.5) | 0.3 (2.4)
  Change at Month 6 | -0.4 (2.4) | 0.4 (2.6)
  Change at Month 9 | -0.2 (2.3) | -0.1 (2.6)
  Change at Month 12 | -0.6 (2.1) | -0.1 (2.6)
Statistical Analysis 1: Comparison: AndroGel® (Testosterone Gel) vs Placebo Gel; Test type: Superiority or Other; p < 0.001, Treatment Effect — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.49, 95% CI 2-sided [-0.79 to -0.19]

17. Secondary Outcome: Vitality Trial - Patient Health Questionnaire 9 (PHQ-9) Change in Overall Score
Description: Baseline score and change in score in the Patient Health Questionnaire 9 (PHQ-9) from baseline to Month 12.
  Scores on the Patient Health Questionnaire 9 (PHQ-9) depression scale range from 0 to 27, with higher scores indicating greater intensity of depressive symptoms.
Time Frame: 1 year (change from baseline to month 3, 6, 9 and 12)
Measure: Mean (Standard Deviation); unit: Score on the PHQ-9 test scale
Arm/Group | AndroGel® (Testosterone Gel) | Placebo Gel
Number analyzed (Participants) | 230 | 234
Score on the PHQ-9 test scale
  Baseline Score | 6.6 (4.0) | 6.6 (4.0)
  Change at Month 3 | -1.3 (3.8) | -0.8 (3.5)
  Change at Month 6 | -1.7 (3.8) | -0.5 (3.7)
  Change at Month 9 | -1.9 (4.0) | -1.2 (4.2)
  Change at Month 12 | -1.8 (3.7) | -1.1 (3.8)
Statistical Analysis 1: Comparison: AndroGel® (Testosterone Gel) vs Placebo Gel; Test type: Superiority or Other; p = 0.004, Treatment Effect — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.72, 95% CI 2-sided [-1.20 to -0.23]

18. Secondary Outcome: Cardiovascular Trial - Total Plaque Volume Change From Baseline
Description: Total plaque volume,mm3 measured by coronary computed tomographic angiography
Time Frame: 1 year (change from baseline to month 12)
Measure: Mean (95% Confidence Interval); unit: mm^3
Arm/Group | AndroGel® (Testosterone Gel) | Placebo Gel
Number analyzed (Participants) | 73 | 65
mm^3 | 75 [22 to 128] | 28 [-24 to 81]
Statistical Analysis 1: Comparison: AndroGel® (Testosterone Gel) vs Placebo Gel; Test type: Superiority; p = .006, Regression, Linear — Determined by linear mixed model with all balancing factors and baseline outcome value as covariates and a random effect for participant; Mean Difference (Final Values) = 47, 95% CI 2-sided [13 to 80] — [estimate comment as in outcome 4, analysis 1]

19. Secondary Outcome: Cardiovascular Trial - Coronary Artery Calcium Score, Agatston Units Change From Baseline
Description: Coronary artery calcium score in Agatston units (range of 0 to >400 Agatston units), with higher values indicating more severe atherosclerosis).
Time Frame: 1 year (change from baseline to month 12)
Population: All participants with measurements of both baseline and 12-month assessments were included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Agatston units
Arm/Group | AndroGel® (Testosterone Gel) | Placebo Gel
Number analyzed (Participants) | 73 | 65
Agatston units | 64 [-19 to 146] | 91 [7 to 174]
Statistical Analysis 1: Comparison: AndroGel® (Testosterone Gel) vs Placebo Gel; Test type: Superiority; p = .31, Regression, Linear — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = -27, 95% CI 2-sided [-80 to 26] — [estimate comment as in outcome 4, analysis 1]

20. Secondary Outcome: Bone Trial - Volumetric Bone Mineral Density (BMD) of Spine Peripheral Bone by Quantitative Computed Tomography (QCT)
Description: Spine peripheral bone as measured by QCT, mg/cm3 (within-arm mean percent change between baseline and month 12 adjusted for balancing factors)
Time Frame: 1 year (baseline to month 12)
Measure: Mean (95% Confidence Interval); unit: percentage of change
Arm/Group | AndroGel® (Testosterone Gel) | Placebo Gel
Number analyzed (Participants) | 110 | 97
percentage of change | 4.0 [2.9 to 5.2] | 1.1 [0.0 to 2.2]
Statistical Analysis 1: Comparison: AndroGel® (Testosterone Gel) vs Placebo Gel; Test type: Superiority; p < .001, Regression, Linear — Treatment effect is the mean difference in the change from baseline between testosterone and placebo arms. The P-Value for the significance of the treatment effect was determined by multivariable linear regression adjusted for balancing factors; Mean Difference (Final Values) = 2.9, 95% CI 2-sided [2.1 to 3.7]

21. Secondary Outcome: Bone Trial - Volumetric Bone Mineral Density (BMD) of Spine Whole Bone by Quantitative Computed Tomography (QCT)
Description: Spine whole bone as measured by QCT, mg/cm3 (within-arm mean percent change between baseline and month 12 adjusted for balancing factors)
Time Frame: 1 year (baseline to month 12)
Measure: Mean (95% Confidence Interval); unit: percentage of change
Arm/Group | AndroGel® (Testosterone Gel) | Placebo Gel
Number analyzed (Participants) | 110 | 97
percentage of change | 5.5 [4.0 to 6.9] | 1.2 [-0.2 to 2.6]
Statistical Analysis 1: Comparison: AndroGel® (Testosterone Gel) vs Placebo Gel; Test type: Superiority; p < .001, Regression, Linear — [p-value comment as in outcome 20, analysis 1]; Mean Difference (Final Values) = 4.2, 95% CI 2-sided [3.2 to 5.3]

22. Secondary Outcome: Bone Trial - Volumetric Bone Mineral Density (BMD) of Hip Trabecular Bone by Quantitative Computed Tomography (QCT)
Description: Hip trabecular bone as measured by QCT, mg/cm3 (within-arm mean percent change between baseline and month 12 adjusted for balancing factors)
Time Frame: 1 year (baseline to month 12)
Measure: Mean (95% Confidence Interval); unit: percentage of change
Arm/Group | AndroGel® (Testosterone Gel) | Placebo Gel
Number analyzed (Participants) | 103 | 88
percentage of change | 1.6 [0.8 to 2.4] | 0.1 [-0.6 to 0.9]
Statistical Analysis 1: Comparison: AndroGel® (Testosterone Gel) vs Placebo Gel; Test type: Superiority; p < .001, Regression, Linear — [p-value comment as in outcome 20, analysis 1]; Median Difference (Final Values) = 1.5, 95% CI 2-sided [0.9 to 2.0]

23. Secondary Outcome: Bone Trial - Volumetric Bone Mineral Density (BMD) of Hip Peripheral Bone by Quantitative Computed Tomography (QCT)
Description: Hip peripheral bone as measured by QCT, mg/cm3 (within-arm mean percent change between baseline and month 12 adjusted for balancing factors)
Time Frame: 1 year (baseline to month 12)
Measure: Mean (95% Confidence Interval); unit: percentage of change
Arm/Group | AndroGel® (Testosterone Gel) | Placebo Gel
Number analyzed (Participants) | 103 | 88
percentage of change | 1.6 [0.9 to 2.3] | 0.7 [-0.0 to 1.4]
Statistical Analysis 1: Comparison: AndroGel® (Testosterone Gel) vs Placebo Gel; Test type: Superiority; p < .001, Regression, Linear — [p-value comment as in outcome 20, analysis 1]; Mean Difference (Final Values) = 1.0, 95% CI 2-sided [0.5 to 1.5]

24. Secondary Outcome: Bone Trial - Volumetric Bone Mineral Density (BMD) of Hip Whole Bone by Quantitative Computed Tomography (QCT)
Description: Hip whole bone as measured by QCT, mg/cm3 (within-arm mean percent change between baseline and month 12 adjusted for balancing factors)
Time Frame: 1 year (baseline to month 12)
Measure: Mean (95% Confidence Interval); unit: percentage of change
Arm/Group | AndroGel® (Testosterone Gel) | Placebo Gel
Number analyzed (Participants) | 103 | 88
percentage of change | 1.7 [1.0 to 2.4] | 0.4 [-0.2 to 1.1]
Statistical Analysis 1: Comparison: AndroGel® (Testosterone Gel) vs Placebo Gel; Treatment effect is the mean difference in the change from baseline between testosterone and placebo arms. The P-Value for the significance of the treatment effect was determined by multivariable linear regression adjusted for balancing factors; Test type: Superiority; p < .001, Regression, Linear; Mean Difference (Final Values) = 1.3, 95% CI 2-sided [0.8 to 1.7]

25. Secondary Outcome: Bone Trial - Bone Strength of Spine Whole Bone by Finite Element Analysis, N
Description: Spine whole bone (within-arm mean percent change between baseline and month 12 adjusted for balancing factors)
Time Frame: 1 year (baseline to month 12)
Measure: Mean (95% Confidence Interval); unit: percentage of change
Arm/Group | AndroGel® (Testosterone Gel) | Placebo Gel
Number analyzed (Participants) | 110 | 97
percentage of change | 9.0 [6.4 to 11.6] | 1.9 [-0.6 to 4.4]
Statistical Analysis 1: Comparison: AndroGel® (Testosterone Gel) vs Placebo Gel; Test type: Superiority; p < .001, Regression, Linear — [p-value comment as in outcome 20, analysis 1]; Mean Difference (Final Values) = 7.1, 95% CI 2-sided [5.3 to 809]

26. Secondary Outcome: Bone Trial - Bone Strength of Spine Trabecular Bone by Finite Element Analysis, N
Description: Spine trabecular bone (within-arm mean percent change between baseline and month 12 adjusted for balancing factors)
Time Frame: 1 year (baseline to month 12)
Measure: Mean (95% Confidence Interval); unit: percentage of change
Arm/Group | AndroGel® (Testosterone Gel) | Placebo Gel
Number analyzed (Participants) | 110 | 97
percentage of change | 10.8 [7.4 to 14.3] | 2.4 [-1.0 to 5.7]
Statistical Analysis 1: Comparison: AndroGel® (Testosterone Gel) vs Placebo Gel; Test type: Superiority; p < .001, Regression, Linear — [p-value comment as in outcome 20, analysis 1]; Mean Difference (Final Values) = 8.5, 95% CI 2-sided [6.0 to 10.9]

27. Secondary Outcome: Bone Trial - Bone Strength of Spine Peripheral Bone by Finite Element Analysis, N
Description: Spine peripheral bone (within-arm mean percent change between baseline and month 12 adjusted for balancing factors)
Time Frame: 1 year (baseline to month 12)
Measure: Mean (95% Confidence Interval); unit: percentage of change
Arm/Group | AndroGel® (Testosterone Gel) | Placebo Gel
Number analyzed (Participants) | 110 | 97
percentage of change | 7.2 [5.2 to 9.2] | 1.5 [-0.5 to 3.4]
Statistical Analysis 1: Comparison: AndroGel® (Testosterone Gel) vs Placebo Gel; Test type: Superiority; p < .001, Regression, Linear — [p-value comment as in outcome 20, analysis 1]; Mean Difference (Final Values) = 5.7, 95% CI 2-sided [4.3 to 7.2]

28. Secondary Outcome: Bone Trial - Bone Strength of Hip Whole Bone by Finite Element Analysis, N
Description: Hip whole bone (within-arm mean percent change between baseline and month 12 adjusted for balancing factors)
Time Frame: 1 year (baseline to month 12)
Measure: Mean (95% Confidence Interval); unit: percentage of change
Arm/Group | AndroGel® (Testosterone Gel) | Placebo Gel
Number analyzed (Participants) | 103 | 88
percentage of change | 2.5 [1.4 to 3.5] | 0.6 [-0.4 to 1.7]
Statistical Analysis 1: Comparison: AndroGel® (Testosterone Gel) vs Placebo Gel; Test type: Superiority; p < .001, Regression, Linear — [p-value comment as in outcome 20, analysis 1]; Mean Difference (Final Values) = 1.8, 95% CI 2-sided [1.1 to 2.6]

29. Secondary Outcome: Bone Trial - Bone Strength of Hip Trabecular Bone by Finite Element Analysis, N
Description: Hip trabecular bone (within-arm mean percent change between baseline and month 12 adjusted for balancing factors)
Time Frame: 1 year (baseline to month 12)
Measure: Mean (95% Confidence Interval); unit: percentage of change
Arm/Group | AndroGel® (Testosterone Gel) | Placebo Gel
Number analyzed (Participants) | 103 | 88
percentage of change | 1.5 [0.5 to 2.5] | 0.5 [-0.5 to 1.5]
Statistical Analysis 1: Comparison: AndroGel® (Testosterone Gel) vs Placebo Gel; Test type: Superiority; p = .005, Regression, Linear — [p-value comment as in outcome 20, analysis 1]; Mean Difference (Final Values) = 1.0, 95% CI 2-sided [0.3 to 1.7]

30. Secondary Outcome: Bone Trial - Bone Strength of Hip Peripheral Bone by Finite Element Analysis, N
Description: Hip peripheral bone (within-arm mean percent change between baseline and month 12 adjusted for balancing factors)
Time Frame: 1 year (baseline to month 12)
Measure: Mean (95% Confidence Interval); unit: percentage of change
Arm/Group | AndroGel® (Testosterone Gel) | Placebo Gel
Number analyzed (Participants) | 103 | 88
percentage of change | 1.4 [0.7 to 2.0] | 0.4 [-0.3 to 1.0]
Statistical Analysis 1: Comparison: AndroGel® (Testosterone Gel); Test type: Superiority; p < .001, Regression, Linear — [p-value comment as in outcome 20, analysis 1]; Mean Difference (Final Values) = 1.0, 95% CI 2-sided [0.5 to 1.4]

31. Secondary Outcome: Bone Trial - Area Bone Mineral Density (BMD) of Lumbar Spine by Dual-energy X-ray Absorptiometry (DXA)
Description: Lumbar spine as measured by DXA, g/cm2 (within-arm mean percent change between baseline and month 12 adjusted for balancing factors)
Time Frame: 1 year (baseline to month 12)
Measure: Mean (95% Confidence Interval); unit: percentage of change
Arm/Group | AndroGel® (Testosterone Gel) | Placebo Gel
Number analyzed (Participants) | 109 | 101
percentage of change | 3.3 [2.01 to 4.56] | 2.1 [0.87 to 3.36]
Statistical Analysis 1: Comparison: AndroGel® (Testosterone Gel) vs Placebo Gel; Test type: Superiority; p = .01, Regression, Linear — [p-value comment as in outcome 20, analysis 1]; Mean Difference (Final Values) = 1.2, 95% CI 2-sided [0.25 to 2.09]

32. Secondary Outcome: Bone Trial - Area Bone Mineral Density (BMD) of Total Hip by Dual-energy X-ray Absorptiometry (DXA)
Description: Total hip as measured by DXA, g/cm2 (within-arm mean percent change between baseline and month 12 adjusted for balancing factors)
Time Frame: 1 year (baseline to month 12)
Measure: Mean (95% Confidence Interval); unit: percentage of change
Arm/Group | AndroGel® (Testosterone Gel) | Placebo Gel
Number analyzed (Participants) | 108 | 100
percentage of change | 1.2 [0.19 to 2.17] | 0.5 [-0.45 to 1.46]
Statistical Analysis 1: Comparison: AndroGel® (Testosterone Gel) vs Placebo Gel; Test type: Superiority; p = .052, Regression, Linear — [p-value comment as in outcome 20, analysis 1]; Mean Difference (Final Values) = .07, 95% CI 2-sided [-0.01 to 1.36]

33. Secondary Outcome: Bone Trial - Area Bone Mineral Density (BMD) of Femoral Neck by Dual-energy X-ray Absorptiometry (DXA)
Description: Femoral neck as measured by DXA, g/cm2 (within-arm mean percent change between baseline and month 12 adjusted for balancing factors)
Time Frame: 1 year (baseline to month 12)
Measure: Mean (95% Confidence Interval); unit: percentage of change
Arm/Group | AndroGel® (Testosterone Gel) | Placebo Gel
Number analyzed (Participants) | 108 | 100
percentage of change | 1.5 [0.02 to 2.97] | 0.9 [-0.49 to 2.35]
Statistical Analysis 1: Comparison: AndroGel® (Testosterone Gel) vs Placebo Gel; Test type: Superiority; p = 0.27, Regression, Linear — [p-value comment as in outcome 20, analysis 1]; Mean Difference (Final Values) = 0.56, 95% CI 2-sided [-0.45 to 1.58]

34. Secondary Outcome: Cognitive Function Trial - Visual Memory - Benton Visual Retention Test (BVRT)
Description: Baseline score and mean change in score in the Visual Memory Using the Benton Visual Retention Test (BVRT) from baseline, Month 6 and Month 12.
  The BVRT measures short term visual memory and visuo-constructional abilities and was administered and scored according to standard procedures. Each of 10 designs was presented one at a time for 10 seconds, and immediately after the design was withdrawn, the participant was instructed to draw it from memory on a blank sheet of paper. The score was the total number of figures with errors and ranged from 0 to 26. Scores were inverted to 0 to -26 so that higher scores would reflect better performance.
  Change in BVRT scores from baseline are treated as continuous and compared between AAMI Androgel and placebo subjects using linear random effects models adjusting for balancing factors as described in the primary analysis.
Time Frame: 1 year (baseline to month 6 and month 12)
Measure: Mean (95% Confidence Interval); unit: Score on the BVRT test scale
Arm/Group | AndroGel® (Testosterone Gel) | Placebo Gel
Number analyzed (Participants) | 246 | 246
Score on the BVRT test scale
  Baseline Score | -8.2 [-8.6 to -7.8] | -8.2 [-8.6 to -7.8]
  Change at Month 6 | 0.2 [-0.4 to 0.9] | 0.3 [-0.3 to 1.0]
  Change at Month 12 | 0.3 [-0.4 to 0.9] | 0.7 [0.0 to 1.4]
Statistical Analysis 1: Comparison: AndroGel® (Testosterone Gel) vs Placebo Gel; A positive estimated difference indicates greater increases, smaller decreases, or both for the testosterone group compared with the placebo group; Test type: Superiority; p = .24, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-0.76 to 0.19] — The difference is the mean difference in the change from baseline to 6 months to 12 months in participants allocated to testosterone vs placebo adjusted for balancing factors

35. Secondary Outcome: Cognitive Function Trial - Spatial Ability Card Rotation Test (CRT)
Description: Baseline score and change in score in the Spatial Ability Using the Card Rotation Test at baseline, Month 6 and Month 12.
  Change in performance on the Card Rotations Test will be analyzed using linear random effects models adjusting for baseline performance, balancing factors, education, and test version. The test consists of a series of 10 primary figures, each of which has 8 corresponding secondary figures. Subjects are asked to determine which of the secondary figures is the same as the corresponding primary figure, and the score is taken as the number of figures answered correctly minus the number of figures answered incorrectly.
  The maximum score is 80 for subjects who answer all items correctly.
Time Frame: 1 year (baseline to month 6 to month 12)
Measure: Mean (95% Confidence Interval); unit: Score on the CRT test scale
Arm/Group | AndroGel® (Testosterone Gel) | Placebo Gel
Number analyzed (Participants) | 245 | 243
Score on the CRT test scale
  Baseline Score | 28.7 [26.9 to 30.5] | 30.0 [28.1 to 31.8]
  Change at Month 6 | 0.6 [-1.9 to 30.] | 0.2 [-2.3 to 2.7]
  Change at Month 12 | 0.6 [-1.8 to 3.1] | 1.2 [-1.3 to 3.7]
Statistical Analysis 1: Comparison: AndroGel® (Testosterone Gel) vs Placebo Gel; [analysis description as in outcome 34, analysis 1]; Test type: Superiority; p = .89, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Net) = -0.12, 95% CI 2-sided [-1.89 to 1.65] — [estimate comment as in outcome 34, analysis 1]

36. Secondary Outcome: Cognitive Function Trial - Executive Function - Trail Making Test B - A
Description: Baseline score and change in score in Executive Function as Measured by Trail-Making Test (TMT) B - A, at baseline, Month 6 and Month 12.
  Change in performance on the Trail Making Test was analyzed using linear random effects models adjusting for baseline performance, balancing factors, education, and test version.
  Participants are required to connect a set of numbers (Part A) or alternating letters and numbers (Part B) in sequential order. The score for each part is the total time (in seconds) to complete both parts. The outcome analyzed will be the total time for Trails B minus the total time for Trails A to provide a measure of working memory, adjusted for attention and processing speed. Higher scores reflect lower executive function.
Time Frame: 1 year (baseline to month 6 to month 12)
Measure: Mean (95% Confidence Interval); unit: Score on the Trail Making Test scale
Arm/Group | AndroGel® (Testosterone Gel) | Placebo Gel
Number analyzed (Participants) | 245 | 245
Score on the Trail Making Test scale
  Baseline Score | 86.4 [78.3 to 94.6] | 76.7 [69.9 to 83.5]
  Change at Month 6 | -2.1 [-12.4 to 8.2] | 1.8 [-8.6 to 12.2]
  Change at Month 12 | -0.0 [-10.3 to 10.3] | 7.1 [-3.3 to 17.5]
Statistical Analysis 1: Comparison: AndroGel® (Testosterone Gel) vs Placebo Gel; [analysis description as in outcome 34, analysis 1]; Test type: Superiority; p = .14, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Net) = -5.51, 95% CI 2-sided [-12.91 to 1.88] — [estimate comment as in outcome 34, analysis 1]

37. Secondary Outcome: Anemia Trial - Effect of Testosterone on Hemoglobin Levels - Unexplained Anemia - Hemoglobin (Continuous)
Description: Proportion of men age 65 years or older with unexplained anemia who increased their hemoglobin level by 1.0 gm/dL from baseline.
  Values are means (SDs) for continuous outcomes.
Time Frame: 1 year (baseline to month 12)
Measure: Mean (Standard Deviation); unit: proportion of participants
Arm/Group | AndroGel® (Testosterone Gel) | Placebo Gel
Number analyzed (Participants) | 27 | 35
proportion of participants | 0.9 (1.4) | 0.2 (0.8)
Statistical Analysis 1: Comparison: AndroGel® (Testosterone Gel) vs Placebo Gel; Test type: Superiority; p < .001, Mixed Models Analysis — The P-value for the significance of the treatment effect was determined by a linear mixed model for continuous outcomes with a random intercept for participant; Mean Difference (Net) = 0.83, 95% CI 2-sided [0.48 to 1.39] — Intent-to-treat analysis by a linear mixed effects model adjusted for balancing factors

ADVERSE EVENTS:
Time Frame: Adverse events were identified during study visits in the First (Treatment) Year, and by phone interview during the Second (Observation) Year.
Description: All adverse events were coded by an independent expert. Cardiovascular adverse events were collected by a specific questionnaire administered at each visit during treatment and for one year after treatment.
  Cardiovascular adverse events were also identified from the Adverse Event log and SAE Report Forms. Cardiovascular events were adjudicated.
  Myocardial infarction, stroke and death were adjudicated by two adjudicators, and all other events by one adjudicator.
Arm/Group | AndroGel® (Testosterone Gel) | Placebo Gel
Serious Adverse Events (participants affected / at risk) | 183/394 | 176/394
Other Adverse Events (participants affected / at risk) | 343/394 | 341/394
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AndroGel® (Testosterone Gel) (N=394) | Placebo Gel (N=394)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Cardiac disorders (Cardiac disorders) | 35 (38) | 34 (42)
Gastrointestinal disorders (Gastrointestinal disorders) | 10 (10) | 7 (8)
Hepatobiliary disorders (Hepatobiliary disorders) | 4 (4) | 2 (3)
Infections and infestations (Infections and infestations) | 29 (34) | 21 (25)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 9 (11) | 11 (14)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 22 (24) | 19 (22)
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15 (16) | 12 (14)
Nervous system disorders (Nervous system disorders) | 16 (17) | 22 (24)
Psychiatric disorders (Psychiatric disorders) | 3 (5) | 1 (1)
Renal and urinary disorders (Renal and urinary disorders) | 4 (5) | 1 (1)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Respiratory disorders (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 17 (22)
Surgical and medical procedures (Surgical and medical procedures) | 1 (1) | 1 (1)
Vascular disorders (Vascular disorders) | 10 (12) | 7 (7)
General disorders (General disorders) | 12 (13) | 14 (15)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AndroGel® (Testosterone Gel) (N=394) | Placebo Gel (N=394)
Cardiac disorders (Cardiac disorders) | 45 (82) | 45 (88)
Infections and infestations (Infections and infestations) | 152 (221) | 145 (220)
Eye disorders (Eye disorders) | 23 (27) | 27 (36)
Gastrointestinal disorders (Gastrointestinal disorders) | 65 (99) | 71 (116)
General disorders and administration site conditions (General disorders) | 74 (115) | 75 (99)
Injury poisoning and procedural complications (Injury, poisoning and procedural complications) | 87 (143) | 89 (160)
Investigations (Investigations) | 45 (59) | 37 (54)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 24 (31) | 29 (34)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 145 (272) | 155 (293)
Neoplasms benign, malignant and unspecified (including cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 28 (35) | 22 (27)
Nervous system disorders (Nervous system disorders) | 75 (101) | 78 (107)
Psychiatric disorders (Psychiatric disorders) | 26 (41) | 27 (37)
Renal and urinary disorders (Renal and urinary disorders) | 43 (59) | 42 (53)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 49 (63) | 19 (22)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 74 (110) | 67 (106)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 88 (156) | 52 (75)
Surgical and medical procedures (Surgical and medical procedures) | 36 (55) | 31 (43)
Vascular disorders (Vascular disorders) | 33 (42) | 34 (43)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No